CLINICAL TRIAL: NCT03932409
Title: A Phase Ib Trial of Vaginal Cuff Brachytherapy + Pembrolizumab (MK3475) Followed by 3 Cycles of Dose Dense Paclitaxel/q 21 Day Carboplatin + Pembrolizumab (MK3475) in High Intermediate Risk Endometrial Cancer
Brief Title: Frontline Immunotherapy Combined With Radiation and Chemotherapy in High Risk Endometrial Cancer
Acronym: FIERCE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-FIERCE
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer
Keywords: pembrolizumab; radiation therapy
MeSH Terms: conditions — Endometrial Neoplasms | interventions — pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Radiation Therapy + Pembrolizumab/Chemotherapy (Experimental): Pembrolizumab given 7 days prior to radiation therapy (e.g., vaginal cuff brachytherapy) followed by three cycles pembrolizumab combined with Carboplatin/Paclitaxel chemotherapy
  Interventions: Drug: Pembrolizumab; Radiation: Vaginal cuff brachytherapy (VCB); Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab — prior to VCB: 200mg IV given one week (7 days) before radiation
  after VCB: 200mg IV on day 1 of a 21 day cycle prior to chemotherapy
  Other Names: MK3475
Radiation: Vaginal cuff brachytherapy (VCB) — Treatment should commence within 12 weeks of the surgery/hysterectomy
Drug: Paclitaxel — after VCB, Paclitaxel IV on days 1,8 and 15 of a 21 day cycle for 3 cycles
Drug: Carboplatin — after VCB, Carboplatin IV on day 1 of a 21 day cycle for 3 cycles

SUMMARY:
The purpose of this single arm, open label study is to evaluate the feasibility of pembrolizumab combined with radiation administered to the upper part of the vagina (vaginal cuff brachytherapy) followed by three cycles of pembrolizumab and chemotherapy in patients with endometrial cancer.

DETAILED DESCRIPTION:
Before the patient begins the study:

Endometrial cancer is commonly treated with surgery. The patient must have already had surgery including hysterectomy (removal of the uterus) prior to being considered eligible for this study. The surgery may also include removal of the ovaries, and removal of pelvic and para-aortic lymph nodes. Following the surgery, the doctor will identify if the patient has factors related to the cancer which places the patient at a greater risk for the cancer returning.

Prior to participating in this study there are exams, tests or procedures to find out if the patient can be treated in the study. Most are part of regular cancer care. Tumor tissue will need to be collected for study tests to see if the patient is eligible for to take part on the study.

TREATMENT If the patient is eligible, pembrolizumab will be given 7 days before radiation therapy. After radiation therapy, three cycles of pembrolizumab and chemotherapy will be given.

Study participation will be up to two years.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have undergone hysterectomy. Bilateral salpingooophorectomy is strongly encouraged but not mandatory.
2. Pelvic and para-aortic lymphadenectomy are optional, but strongly encouraged.
3. If either a bilateral salpingo-oophorectomy (BSO) or nodal sampling was not performed, post-operative pre-treatment CT/MRI is required and must not demonstrate evidence suggestive of metastatic disease (adnexa, nodes, intraperitoneal disease). Post-operative, pre-treatment CT/MRI must be performed if a BSO and/or lymphnode sampling was not performed.
4. Tissue from an archival sample or newly obtained core or excisional biopsy of a tumor lesion within 10 weeks confirming diagnosis.
5. All patients will be staged according to the FIGO 2009 staging system and with endometrial carcinoma (endometrioid types) confined to the corpus uteri or with endocervical glandular involvement fitting one of the following high-intermediate risk factor categories:

   * age ≥18 years with 3 risk factors
   * Risk factors:

     1. Grade 2 or 3 tumor, (+) lymphovascular space invasion, outer ½ myometrial invasion. Patients with these risk criteria may be enrolled with either positive or negative cytology.
     2. Patients with Stage II endometrial carcinoma (any histology) with cervical stromal invasion (occult or gross involvement), with or without high-intermediate risk factors.
     3. Patients with serous or clear cell histology (with or without other high-intermediate risk factors) are eligible provided the disease is Stage I or II (with or without cervical stromal invasion or endocervical glandular involvement). Eligibility for clear cell and serous histology is not based on presence of lymphovascular space invasion or depth of invasion.
6. Patients must have ECOG performance status 0 or 1.
7. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial and authorization permitting release of personal health information.
8. Neuropathy (sensory and motor) ≤ Grade 1.
9. Have adequate organ function as defined per Protocol.

Exclusion Criteria:

1. Patients with recurrent disease.
2. Greater than 12 weeks elapsed from surgery to enrollment
3. Patients have prior pelvic or abdominal radiation therapy
4. Known hypersensitivity to any component of study treatments that resulted in drug discontinuation
5. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
6. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to allocation.
7. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
8. Has received a live vaccine within 30 days prior to the first dose of study drug.
9. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
12. Has known active CNS metastases and/or carcinomatous meningitis.
13. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
16. Has an active infection requiring systemic therapy. This excludes grade 2 urinary tract infections or grade 1-2 skin infections.
17. Has a known history of Human Immunodeficiency Virus (HIV).
18. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
19. Has a known history of active TB (Bacillus Tuberculosis).
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Is pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients completing three cycles | 4 months
  defined as completion of 3 cycles of pembrolizumab combined with dose dense paclitaxel and carboplatin chemotherapy

SECONDARY OUTCOMES:
progression free survival | up to 2 years
  time from study entry to the first tumor progression
progression free survival | 6 months
  progression free survival rate at 6 months
Overall survival | up to 2 years
  time from study entry to death
Frequency of adverse events | 5 months
  frequency and severity of adverse events as assessed by the CTCAE v5

CONTACTS AND LOCATIONS:
Overall Officials: Christina Washington, MD, Principal Investigator — Stephenson Cancer Center
Locations (2):
- United States (2):
  - LSU Health New Orleans, New Orleans, Louisiana
  - Stephenson Cancer Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No